CLINICAL TRIAL: NCT06753513
Title: Clinical Application of 99mTc-FDPH46 SPECT/CT Imaging in Malignant Solid Tumor: a Prospective Exploratory Study
Acronym: 99mTc；FAPI；mCi
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhang jun, Deputy Chief Physician, Zhejiang University
Other Study IDs: IIT20240134C-R1
Record Dates: First submitted 2024-12-10; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Malignant Tumors; Solid Tumor Malignancy
Keywords: 99mTc; FDPH46; SPECT; Malignant Solid Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient Self-Control: Patient Self-Control
  Interventions: Other: 99mTc-FDPH46 SPECT/CT Imaging

INTERVENTIONS:
Other: 99mTc-FDPH46 SPECT/CT Imaging — 99mTc-FDPH46 SPECT/CT Imaging

SUMMARY:
The goal of this observational study aims to preliminarily evaluate the diagnostic efficacy of 99mTc-FDPH46 SPECT/CT in malignant solid tumors (compared to the pathological gold standard). The main questions it aims to answer are:

* What is the diagnostic efficacy of 99mTc-FDPH46 in malignant solid tumors, compared to the pathological gold standard?
* What is the biodistribution, tumor uptake and safety of 99mTc-FDPH46 SPECT/CT in patients with malignant solid tumors?

Participant Will:

• Patients with clinically suspected or diagnosed malignant solid tumors who are willing to undergo 99mTc-FDPH46 SPECT/CT examination and sign an informed consent form.

DETAILED DESCRIPTION:
Patients who are clinically assessed as suspected or diagnosed with malignant solid tumors will receive an intravenous injection of 20-25mCi of 99mTc-FDPH46. Whole-body planar scintigraphy will be performed at 10, 30, 90, 150, and 240 minutes post-injection to obtain dynamic biodistribution images. Additionally, 99mTc-FDPH46 SPECT/CT imaging will be conducted 60-90 minutes after the intravenous injection to acquire both whole-body planar scintigraphy and SPECT/CT tomographic fusion images. After the scans are completed, patients will be observed in the waiting room for 1 hour before they are allowed to return.During the follow-up visit after the examination, the researchers will collect the patients' clinical information and any changes in symptoms, and record them in the medical records. All subjects will be followed up once on the same day after the SPECT/CT scan and again one week later.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are clinically suspected or diagnosed with malignant solid tumors.
2. Ages between 18 to 80 years old.
3. Stable vital signs, ECOG score of 0-2, capable of tolerating and cooperating with the 99mTc-FDPH46 SPECT/CT examination.
4. Subjects who are willing to undergo the 99mTc-FDPH46 SPECT/CT examination and have signed the informed consent form.

Exclusion Criteria:

1. Those who can not understand, comply with the research protocol or are unable to sign the informed consent form.
2. Contraindications for SPECT imaging (including pregnant women, nursing women, women of childbearing age with recent plans to conceive, etc.).
3. Unstable vital signs, ECOG score >2, unable to tolerate or cooperate with the 99mTc-FDPH46 SPECT/CT examination process.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are clinically suspected or diagnosed with malignant solid tumors.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-28 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compared with the pathological gold standard, assess the diagnostic efficacy of 99mTc-FDPH46 in malignant solid tumors. | 2024.12-2026.10
  Using the pathological gold standard as a reference, the sensitivity, specificity, positive predictive value, and negative predictive value of 99mTc-FDPH46 in patients with malignant solid tumors were evaluated. The consistency between the two diagnostic methods was assessed by Kappa analysis, thereby determining the diagnostic efficacy of 99mTc-FDPH46 in patients with malignant solid tumors.

SECONDARY OUTCOMES:
Assess the safety, biodistribution, and tumor uptake of 99mTc-FDPH46 SPECT/CT in patients with malignant solid tumors. | 2024.12-2026.12
  Assess the safety of 99mTc-FDPH46 SPECT/CT in patients with malignant solid tumors, recording any adverse reactions such as nausea, vomiting, and damage to liver and kidney functions; meanwhile, use the standardized uptake value (SUV) for a quantitative analysis of the tracer's biodistribution and tumor uptake in the patients' bodies.

CONTACTS AND LOCATIONS:
Locations (1):
- No. 79, Qingchun Road, Shangcheng District, Hangzhou City, Zhejiang Province, China., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruan Q, Feng J, Jiang Y, Zhang X, Duan X, Wang Q, Yin G, Xiao D, Zhang J. Preparation and Bioevaluation of 99mTc-Labeled FAP Inhibitors as Tumor Radiotracers to Target the Fibroblast Activation Protein. Mol Pharm. 2022 Jan 3;19(1):160-171. doi: 10.1021/acs.molpharmaceut.1c00712. Epub 2021 Dec 14. PMID 34904839
- [Background] Ruan Q, Zhou C, Wang Q, Kang F, Jiang Y, Li G, Feng J, Zong S, Zhang J, Wang J. A Simple Kit Formulation for Preparation and Exploratory Human Studies of a Novel 99mTc-Labeled Fibroblast Activation Protein Inhibitor Tracer for Imaging of the Fibroblast Activation Protein in Cancers. Mol Pharm. 2023 Jun 5;20(6):2942-2950. doi: 10.1021/acs.molpharmaceut.2c01094. Epub 2023 Apr 21. PMID 37083360
- [Background] Ruan Q, Wang Q, Jiang Y, Feng J, Yin G, Zhang J. Synthesis and Evaluation of 99mTc-Labeled FAP Inhibitors with Different Linkers for Imaging of Fibroblast Activation Proteins in Tumors. J Med Chem. 2023 Apr 13;66(7):4952-4960. doi: 10.1021/acs.jmedchem.2c02062. Epub 2023 Mar 27. PMID 36972467
- [Background] Ruan Q, Ding D, Diao L, Feng J, Yin G, Jiang Y, Wang Q, Han P, Jiang J, Zhang J. Synthesis and Preclinical Evaluation of Novel 99mTc-Labeled FAPI-46 Derivatives with Significant Tumor Uptake and Improved Tumor-to-Nontarget Ratios. J Med Chem. 2024 Feb 22;67(4):3190-3202. doi: 10.1021/acs.jmedchem.4c00031. Epub 2024 Feb 6. PMID 38320123
- [Background] Lindner T, Altmann A, Kramer S, Kleist C, Loktev A, Kratochwil C, Giesel F, Mier W, Marme F, Debus J, Haberkorn U. Design and Development of 99mTc-Labeled FAPI Tracers for SPECT Imaging and 188Re Therapy. J Nucl Med. 2020 Oct;61(10):1507-1513. doi: 10.2967/jnumed.119.239731. Epub 2020 Mar 13. PMID 32169911
- [Background] Liu Y, Zhang Q, Zhang Y, Wang J, Wu Y, Yang G, Shi J, Wang F, Xu Z, Jing H. 99mTc-Labeled FAPI SPECT Imaging in Idiopathic Pulmonary Fibrosis: Preliminary Results. Pharmaceuticals (Basel). 2023 Oct 9;16(10):1434. doi: 10.3390/ph16101434. PMID 37895905
- [Background] Luo X, Zhang Z, Cheng C, Wang T, Fang D, Zuo C, Yuan G, Li R, Li X. SPECT Imaging with Tc-99m-Labeled HYNIC-FAPI-04 to Extend the Differential Time Window in Evaluating Tumor Fibrosis. Pharmaceuticals (Basel). 2023 Mar 10;16(3):423. doi: 10.3390/ph16030423. PMID 36986521
- [Background] Jiang Y, Tian Y, Feng B, Zhao T, Du L, Yu X, Zhao Q. A novel molecular imaging probe [99mTc]Tc-HYNIC-FAPI targeting cancer-associated fibroblasts. Sci Rep. 2023 Mar 6;13(1):3700. doi: 10.1038/s41598-023-30806-6. PMID 36879039
- [Background] Ma M, Yang G, Zhao M, Liu Y, Ge X, Jia B, Gao S. Synthesis and Preliminary Study of 99mTc-Labeled HYNIC-FAPi for Imaging of Fibroblast Activation Proteins in Tumors. Mol Pharm. 2024 Feb 5;21(2):735-744. doi: 10.1021/acs.molpharmaceut.3c00886. Epub 2024 Jan 9. PMID 38193393
- [Background] Jia X, Li X, Jia B, Yang Y, Wang Y, Liu Y, Ji T, Xie X, Yao Y, Qiu G, Deng H, Zhu Z, Chen S, Yang A, Gao R. The role of [99mTc]Tc-HFAPi SPECT/CT in patients with malignancies of digestive system: first clinical experience. Eur J Nucl Med Mol Imaging. 2023 Mar;50(4):1228-1239. doi: 10.1007/s00259-022-06068-1. Epub 2022 Dec 7. PMID 36477400
- [Background] Trujillo-Benitez D, Luna-Gutierrez M, Ferro-Flores G, Ocampo-Garcia B, Santos-Cuevas C, Bravo-Villegas G, Morales-Avila E, Cruz-Nova P, Diaz-Nieto L, Garcia-Quiroz J, Azorin-Vega E, Rosato A, Melendez-Alafort L. Design, Synthesis and Preclinical Assessment of 99mTc-iFAP for In Vivo Fibroblast Activation Protein (FAP) Imaging. Molecules. 2022 Jan 1;27(1):264. doi: 10.3390/molecules27010264. PMID 35011496
- [Background] Boschi A, Urso L, Uccelli L, Martini P, Filippi L. 99mTc-labeled FAPI compounds for cancer and inflammation: from radiochemistry to the first clinical applications. EJNMMI Radiopharm Chem. 2024 May 2;9(1):36. doi: 10.1186/s41181-024-00264-0. PMID 38695960